CLINICAL TRIAL: NCT00283322
Title: Heparin Antibodies in Intensive Care Unit Patients (HAICU)
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Robert L. Levine, MD, The University of Texas Health Science Center at Houston
Other Study IDs: HSC-MS-04-0312; HAICU
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Heparin-Induced Thrombocytopenia
Keywords: Heparin Induced Thrombocytopenia; HIT; HITT; Thrombosis; Thromboembolism
MeSH Terms: conditions — Thrombosis; Thromboembolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma. Patients consented for use to look for heparin antibodies in this study only.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Medical ICU patients: Patients admitted to a medical intensive care unit
  Interventions: Other: blood samples (2)
- Surgical ICU patients: Patients admitted to a surgical-trauma intensive care unit
  Interventions: Other: blood samples (2)
- Neuro ICU patients: Patients admitted to a neuro-trauma intensive care unit
  Interventions: Other: blood samples (2)

INTERVENTIONS:
Other: blood samples (2) — Two blood samples were obtained from patients and tested for heparin antibodies.

SUMMARY:
Intensive care unit patients have multiple risk factors for venous thromboembolism. Venous thromboembolism leads to significant morbidity and can be fatal. Unfractionated heparin and low molecular weight heparin are commonly used to prevent venous thromboembolism. Heparin induced thrombocytopenia, an untoward consequence of exposure to heparin, is an immune disorder that may develop in patients treated with heparin products. Determining the prevalence of heparin induced thrombocytopenia and its relationship to preventive and therapeutic heparin and low molecular weight heparin will help clinicians more appropriately choose methods of venous thromboembolism prophylaxis and treatment in the critically ill, ICU population.

The objective of this study is to determine the prevalence of heparin-induced antibodies on admission to the ICU and the development of new heparin-antibodies during the first week of hospitalization.

DETAILED DESCRIPTION:
Venous Thromboembolism (VTE) is common in the intensive care unit (ICU); VTE leads to significant morbidity and is fatal in 30% of undiagnosed pulmonary emboli and 8% when PE is appropriately treated. Intensive care unit (ICU) patients have multiple risk factors for VTE and tend to be at higher risk than non-ICU patients. Risk factors specific to ICU patients include immobility, central venous catheters, sepsis or infection, need for vasopressors, mechanical ventilation, surgery, trauma, and increasing age. Guidelines exist for the prevention of VTE, and VTE prophylaxis is strongly recommended. Given the high rate of VTE and the attendant morbidity and mortality, most ICU's routinely provide VTE prophylaxis which is individualized according to risk-benefit analysis with respect to thrombosis and bleeding risk. Prophylaxis for patients at risk of bleeding is accomplished by using mechanical compression devices while those without bleeding risk are administered medical prophylaxis which is felt to be more effective.

Recently, it has become apparent that medical prophylaxis is not without risk and that the risk-benefit analysis should also include the risk of developing heparin induced thrombocytopenia (HIT) or heparin induced thrombocytopenia with thrombosis (HITT).

Unfractionated heparin (UFH) and low molecular weight heparin (LMWH) are commonly used to prevent VTE in ICU and non-ICU patients. HIT, an untoward consequence of exposure to heparin is an immune disorder that may develop in patients treated with heparin products. HIT is antibody mediated, usually due to IgG antibodies directed against epitopes on the platelet surface comprised of the heparin-platelet factor 4 complex. HIT is generally characterized by a decrease in platelet count to less than 100 X 109/L, or a 50% decrease from baseline, after exposure to heparin. HIT is typically observed after 5 to 10 days of treatment. Alternatively, patients with previous exposure to heparin can develop HIT in two days while heparin naive patients may develop HIT in about 10 days. The platelet count usually returns to normal several days after discontinuing heparin with or without therapy, though the risk for thrombosis persists for up to 3 months due to the persistence of antibodies.

Using an ELISA assay heparin-induced antibody formation is found in up to 50% of patients exposed to UFH. However, the serotonin release assay (SRA) which is believed to be more specific for HIT detects antibody formation in about 20% of patients. Five percent of patients receiving UFH develop thrombocytopenia (HIT) and half of these patients go on to develop heparin induced thrombocytopenia with thrombosis (HITT) which results in venous and arterial complications which can be life threatening, or result in loss of extremities.

The occurrence of HIT varies widely between clinical populations and is dependent on the type of heparin used, i.e. UFH vs. LMWH. The highest incidence reported to date has been in the cardiac and orthopedic populations and is unknown in the ICU population. Warkentin, et al found in a study of 655 hip surgery patients that 2.7% randomized to UFH developed HIT while none receiving enoxaparin (LMWH) developed HIT. This variability in development of antibodies and the HIT syndrome makes it critically important to understand heparin induced antibody formation as a precursor to HIT and HITT.

Determining the prevalence of HIT and its relationship to preventive and therapeutic UFH and LMWH will help clinicians more appropriately choose methods of VTE prophylaxis and treatment in the critically ill, ICU population.

Objectives To determine the prevalence of heparin-induced antibodies on admission to the ICU and the development of new heparin-antibodies during the first 7 +/- 2 days of hospitalization. Secondary objectives include: determining the incidence of heparin antibody formation in patients treated with UFH, LMWH and mechanical prophylaxis (MPX); and to compare the incidence of heparin antibodies between different ICU populations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years of age) admitted to the

  * Neuro-trauma intensive care unit (NTICU)
  * Shock-trauma intensive care unit (STICU) or
  * Medical intensive care unit (MICU).
* Completed informed consent process.

Exclusion Criteria:

* Admitted to ICU for short-term observation or expected hospital length of stay of less than 5 days
* Undergoing or planned plasmaphoresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive consenting patients admitted to neurotrauma, surgical-trauma or medical intensive care unit meeting enrollment criteria.
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2004-11; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Levine, MD, Principal Investigator — The University of Texas, Houston
Locations (2):
- United States (2):
  - Florida Hospital Center for Hemostasis & Thrombosis (Laboratory), Orlando, Florida
  - UT-Houston/Memorial Hermann Hospital, Houston, Texas